CLINICAL TRIAL: NCT06858423
Title: Budesonide Nasal Irrigation Versus Fluticasone Propionate Nasal Spray in the Treatment of Adult Patients With Allergic Rhinitis
Brief Title: Budesonide Nasal Irrigation Versus Fluticasone Propionate Nasal Spray in Treating Allergic Rhinitis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Eslam Farid Abu Shady ,MD, Lecturer and consultant of otolaryngology, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS-8-8-2023
Record Dates: First submitted 2025-02-14; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Nasal Allergy
Keywords: allergic rhinitis; Budesonide; luticasone propionate
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Sodium Chloride; Nasal Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Saline Group) (Placebo Comparator): 120 patients used 0.9% saline for nasal irrigation.
  Interventions: Other: 0.9% saline for nasal irrigation.
- Group B (Fluticasone Propionate Nasal Spray) (Experimental): 120 patients received fluticasone propionate nasal spray.
  Interventions: Drug: Fluticasone propionate nasal spray.
- Group C (Budesonide Nasal Irrigation) (Experimental): 120 patients received budesonide buffered with 0.9% isotonic saline.
  Interventions: Drug: Budesonide buffered with 0.9% isotonic saline.

INTERVENTIONS:
Drug: Budesonide buffered with 0.9% isotonic saline. — 120 patients received budesonide buffered with 0.9% isotonic saline.
  Arms: Group C (Budesonide Nasal Irrigation)
Drug: Fluticasone propionate nasal spray. — 120 patients received fluticasone propionate nasal spray.
  Arms: Group B (Fluticasone Propionate Nasal Spray)
Other: 0.9% saline for nasal irrigation. — 120 patients used 0.9% saline for nasal irrigation.
  Arms: Group A (Saline Group)

SUMMARY:
Budesonide is a medication of the corticosteroid type. Available as an inhaler, nebulization solution, The inhaled form is used in the long-term management of asthma and chronic obstructive pulmonary disease is used for allergic rhinitis and nasal polyps fluticasone propionate

DETAILED DESCRIPTION:
The current study aims to compare between results of budesonid nasal irrigation and fluticasone nasal spray in the treatment of adult patients with Allergic Rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Adult age between 18 and 60 years old.
* Patients with allergic rhinitis evidence by past skin prick testing. Patients were given a skin prick test with a panel of dog, cat, Dermatophagoides farinae, D pteronyssinus, Alternaria, Penicillium, Hormodendron, Aspergillus, grass pollen mix, tree pollen mix, and ragweed allergen extracts (100,000 Allergen Unit/mL). Histamine, 10 mg/mL, was used as a positive control, and the diluent was used as the negative control. A positive reaction was defined as a wheal diameter at least 3 mm greater than the diluent control and/or at least a 50-mm flare (ie, erythema measured as the sum of the greatest diameter and the perpendicular diameter through the midpoint of the greatest diameter)

Exclusion Criteria:

* Patients who had autoimmune diseases or any immune compromised diseases including diabetes, chemotherapy.
* Patients with a history of nasal surgery.
* Patients who received systemic or topical corticosteroids, herbal drugs, beta blocking agent within the previous month of enrolment.
* Patients with asthma and COPD, nasal bleeding, obstructing nasal polyps, paranasal sinus.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | 1 month
  improvement measured by pre- and post-treatment SNOT score

SECONDARY OUTCOMES:
Endoscopic examination improvement | 1 month
  by comparing pre and post treatment lund*Mackay score

OTHER OUTCOMES:
Effects on serum cortisol level | 1 month
  Monitoring of pre and post treatment measurements of e morning serum cortisol level

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospitals - Otolaryngology department, Banhā, Qalyobia, Egypt

IPD SHARING:
Plan to Share IPD: No